CLINICAL TRIAL: NCT05197660
Title: Routine Surgical Procedures During COVID-19 Pandemic: a French Nationwide Cohort Study
Status: Completed | Type: Observational
Sponsor: EPI-PHARE (Other Government)
Responsible Party: Principal Investigator, Emmanuelle Dufour, pharmacoepidemiologist, French National Agency for Medicines and Health Products Safety, French National Health Insurance, EPI-PHARE
Other Study IDs: EP-0275
Record Dates: First submitted 2022-01-14; First posted 2022-01-19 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Surgery; Cataract; Hip Arthroplasty; Knee Arthroplasty; Coronary Stent; Pacemaker; COVID-19 Pandemic
MeSH Terms: conditions — Cataract; COVID-19 | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- - cataract surgery
  Interventions: Procedure: surgical procedures
- - hip arthoplasty
  Interventions: Procedure: surgical procedures
- - knee arthoplasty
  Interventions: Procedure: surgical procedures
- - coronary angioplasty
  Interventions: Procedure: surgical procedures
- - definitive cardiac stimulation (pacemaker)
  Interventions: Procedure: surgical procedures

INTERVENTIONS:
Procedure: surgical procedures — number of hospital stays

SUMMARY:
Determine the consequences of COVID-19 pandemic on routine targeted surgeries.

Five surgical procedures were considered : cataract surgery, hip and knee arthoplasties, coronary revascularisation by angioplasty and definitive cardiac stimulation.

The objective of the study is to quantify changes of these procedures in 2020 and in 2021 (up to June) compared to 2019 taking into account their annual evolution and according to the type of operation (primary or reoperation/revision) and emergency status, if applicable.

ELIGIBILITY:
Inclusion Criteria:

* hospitalizations with at least one act of cataract surgey hip arthroplasty knee arthroplasty coronary angioplasty definitive cardiac stimulation (pacemaker)
* between January 1, 2019, and June 30, 2021

Exclusion Criteria:

-hospitalizations for personal identifier problems in the database

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All hospitalizations with at least one act of each surgery between January 1, 2019, and June 30, 2021 from the French National Health Data System (SNDS).
  The National Health Data System (SNDS) is a set of strictly anonymous databases, comprising all mandatory national health insurance reimbursement data, particularly data derived from processing of health care claims (electronic or paper claims) and data from health care facilities (PMSI).
Sampling Method: Non-Probability Sample
Enrollment: 2000000 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
observed and expected number | 2020 and first half of 2021

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Zureik, Study Director — EPI-PHARE
Locations (1):
- E Dufour, Saint-Denis, Île-de-France Region, France